CLINICAL TRIAL: NCT01011114
Title: Using Cinacalcet to Treat the Hypophosphatemia of Early Kidney Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not renewed with the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-07-203
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hypophosphatemia; Renal Transplant
Keywords: hypophosphatemia; hyperparathyroidism; renal transplant
MeSH Terms: conditions — Hypophosphatemia; Hyperparathyroidism | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cincalcet (Active Comparator): cinacalcet will be titrated as needed to achieve serum phosphorus of > 2.5 mg/dl randomized, placebo-controlled trial comparing the effect of cinacalcet to placebo in controlling serum phosphorus. All subjects will receive oral phosphorus supplementation and Vitamin D as needed to maintain baseline Phosphorus at ~ 2.5 mg/l.
  Interventions: Drug: Cinacalcet
- Control (Placebo Comparator): subjects will receive placebo pill titrated as needed to achieve phosphorus > 2.5 mg/dl.
  randomized, placebo-controlled trial comparing the effect of cinacalcet to placebo in controlling serum phosphorus. All subjects will receive oral phosphorus supplementation and Vitamin D as needed to maintain baseline Phosphorus at ~ 2.5 mEq/l.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — cinacalcet, 30 mg daily, titrated to achieve serum phosphorus of 2.5 mg/dl, versus placebo, similarly titrated.
  Other Names: Sensipar
  Arms: Cincalcet
Drug: Placebo — cinacalcet, 30 mg daily, titrated to achieve serum phosphorus of 2.5 mg/dl, versus placebo, similarly titrated.
  Arms: Control

SUMMARY:
The purpose of the study is to determine whether cinacalcet, used in patients with secondary hyperparathyroidism to control excessive parathyroid hormone, can normalize low blood phosphorus that is commonly seen in patients who have had a kidney transplant.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (SHPT), common in ESRD, persists following renal transplantation resulting in profound hypophosphatemia. This can lead to hemolysis, congestive heart failure, rhabdomyolysis. Phosphate repletion is difficult in view of the persistent SHPT: oral phosphate supplementation can lead to hypocalcemia, reduced 1,25-OH Vitamin D production, hypercalcemia and further hyperparathyroidism. In addition, phospho-soda has been associated with phosphate nephropathy and renal failure.

Cinacalcet HCl is a calcimimetic agent that has recently become a standard therapy in the treatment of SHPT in ESRD. It suppresses PTH secretion by acting as a modulator of the Calcium-sensing receptor on the PTH cell, causing the PTH cell to decrease production of parathyroid hormone. It is a very effective agent, producing significant reduction of PTH as well as improvement in calcium and phosphate metabolism in the dialysis patient. The drug is well-tolerated with minimal adverse effects. Cinacalcet has also been used to control hypercalcemia in renal transplant patients with persistent hyperparathyroidism. Short-term cinacalcet given for 2 to 4 weeks has normalized serum phosphorus and decreased urinary phosphate wasting in renal transplant recipients with stable graft function.

We hypothesize that Cinacalcet HCl will normalize the hypophosphatemia of early renal transplant by reducing the effects of PTH on the proximal renal tubular transport of phosphorus, thereby allowing phosphate reabsorption and decreasing urinary phosphate wasting.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant within last 3 months
* serum phosphorus less than 2.0 mg/dl
* serum creatinine less than 2.0 mg/dl

Exclusion Criteria:

* sensitivity to cinacalcet
* use of amitryptiline, desipramine, itraconazole, ketoconazole
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2015-10-15 (Actual); Study Completion 2015-10-15 (Actual)

PRIMARY OUTCOMES:
improvement in serum phosphorus | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Coco, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States